CLINICAL TRIAL: NCT01222585
Title: Safety and Pharmacokinetics of Multiple Dose Metronidazole in Premature Infants
Brief Title: Metronidazole Pharmacokinetics (PK) in Premature Infants
Acronym: PTN_METRO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Cohen-Wolkowiez (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, Michael Cohen-Wolkowiez, Assistant Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00024571; HHSN27500003I (Other Grant/Funding Number: NICHD)
Record Dates: First submitted 2010-10-06; First posted 2010-10-18 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-01

CONDITIONS: Serious Systemic Infections; Necrotizing Enterocolitis
Keywords: Metronidazole; Neonate; Premature; Sepsis; Necrotizing enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth; Sepsis | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Intravenous metronidazole loading dose 15 mg/kg followed by 7.5 mg/kg every 12-24 hours
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — Metronidazole will be administered intravenously to premature infants as a 15 mg/kg loading dose followed by maintenance doses of 7.5 mg/kg every 12 hours for infants with >=14 postnatal days and every 24 hours for infants <14 postnatal days.
  Other Names: Flagyl

SUMMARY:
Yearly in the United States over 500,000 newborns are delivered prematurely. This population is at high risk of catastrophic bowel disease known as necrotizing enterocolitis. Infants with necrotizing enterocolitis are at high risk of death, and survivors are at increased risk of mental retardation. Metronidazole is an antibiotic that is often administered to infants with suspected or confirmed necrotizing enterocolitis. Unfortunately, the appropriate dose of metronidazole in premature infants has not been established and it is likely to be different from older children and adults.

The investigators will investigate the appropriate metronidazole dose in very premature infants by: 1) determining how premature infants eliminate metronidazole from the body and 2) determining the safest and most effective dose of metronidazole in premature infants.

The investigators hypothesis are: 1) The rate of removal of metronidazole will increase with infant maturity and 2) an appropriate metronidazole dosing regimen will result in necessary drug levels to treat bacteria involved in necrotizing enterocolitis.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <32 weeks at the time of enrollment.
* Postnatal age <91 days at the time of enrollment.
* Sufficient venous access to permit administration of study medication.
* Infant suspected to have a serious infection and from whom a blood culture has been obtained within 96 hours of study entry.

Exclusion Criteria:

* History of anaphylaxis to metronidazole or other nitroimidazole derivatives (e.g., tinidazole).
* Previous exposure to metronidazole in the week prior to study.
* Previous participation in the study.

Max Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cohen-wolkowiez, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - CHOC Children's, Orange, California
  - Wesely Medical Center, Wichita, Kansas
  - Duke University, Durham, North Carolina

REFERENCES:
- [Result] Cohen-Wolkowiez M, Sampson M, Bloom BT, Arrieta A, Wynn JL, Martz K, Harper B, Kearns GL, Capparelli EV, Siegel D, Benjamin DK Jr, Smith PB; Best Pharmaceuticals for Children Act-Pediatric Trials Network. Determining population and developmental pharmacokinetics of metronidazole using plasma and dried blood spot samples from premature infants. Pediatr Infect Dis J. 2013 Sep;32(9):956-61. doi: 10.1097/INF.0b013e3182947cf8. PMID 23587979

RESULTS

PARTICIPANT FLOW:
Groups:
- Metronidazole IV: Intravenous metronidazole loading dose 15 mg/kg followed by 7.5 mg/kg every 12-24 hours
Period: Overall Study
Arm/Group | Metronidazole IV
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: days] — Post Natal Age (Days)
  days | 27 [1 to 82]
Age, Continuous [Mean (Full Range); unit: weeks] — Gestational age (weeks)
  weeks | 25 [23 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
Birth Weight [Median (Full Range); unit: grams] | 740 [431 to 1466]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve at Steady State
Description: Area under the curve at steady state (AUCss)
Time Frame: pre-dose: 30 min; post-dose:10 min, 3-4,6-8, 12-13, 24-25, 36-37, 48-49, 72-73 hours post dose
Population: The PK analysis was conducted using samples from 23 subjects. One subject died soon after the loading dose and was excluded from the analysis. Two subjects had no multiple dose samples. Thus data from 20 subjects were used to estimate this PK parameter.
Measure: Median (Full Range); unit: mg*hr/L
Arm/Group | Metronidazole IV
Number analyzed (Participants) | 20
mg*hr/L | 178.0 [66.0 to 472.0]

2. Primary Outcome: Loading Dose Maximum Concentration
Description: Loading Dose Maximum concentration (Cmax)
Time Frame: 2-5 days of study drug administration
Population: The sample size contains the number of subjects that had the sample of interest collected.
Measure: Median (Full Range); unit: mg/L
Arm/Group | Metronidazole IV
Number analyzed (Participants) | 19
mg/L | 16.54 [9.18 to 19.63]

3. Primary Outcome: Loading Dose Minimum Concentration
Description: Loading Dose Minimum Concentration (mg/L)
Time Frame: 2-5 days of study drug administration
Population: The sample size contains the number of subjects that had the sample of interest collected.
Measure: Median (Full Range); unit: mg/L
Arm/Group | Metronidazole IV
Number analyzed (Participants) | 17
mg/L | 9.20 [3.21 to 12.82]

4. Primary Outcome: Multiple Dose Maximum Concentration
Description: Multiple Dose Maximum Concentration (mg/L)
Time Frame: 2-5 days of study drug administration
Population: The PK analysis was conducted using samples from 23 subjects. One subject died soon after the loading dose and was excluded from the analysis. Two subjects had no multiple dose samples. Thus data from 20 subjects were used to estimate the multiple dose PK parameter.
Measure: Median (Full Range); unit: mg/L
Arm/Group | Metronidazole IV
Number analyzed (Participants) | 20
mg/L | 16.51 [8.71 to 34.05]

5. Primary Outcome: Multiple Dose Minimum Concentration
Description: Multiple Dose Minimum Concentration (mg/L)
Time Frame: 2-5 days of study drug administration
Population: The sample size contains the number of subjects that had the sample of interest collected.
Measure: Median (Full Range); unit: mg/L
Arm/Group | Metronidazole IV
Number analyzed (Participants) | 21
mg/L | 11.62 [1.29 to 27.05]

6. Primary Outcome: Clearance
Description: Clearance (L/h/kg)
Time Frame: 2-5 days of study drug administration
Population: The PK analysis was conducted using samples from 23 subjects. One subject died soon after the loading dose and was excluded from the analysis. Two subjects had no multiple dose samples. Thus data from 20 subjects were used to estimate the PK parameter.
Measure: Median (Full Range); unit: L/h/kg
Arm/Group | Metronidazole IV
Number analyzed (Participants) | 20
L/h/kg | 0.043 [0.016 to 0.105]

7. Primary Outcome: Volume of Distribution
Description: Volume of Distribution (L/kg)
Time Frame: 2-5 days of study drug administration
Population: as for outcome 6
Measure: Median (Full Range); unit: L/kg
Arm/Group | Metronidazole IV
Number analyzed (Participants) | 20
L/kg | 0.99 [0.38 to 2.67]

ADVERSE EVENTS:
Time Frame: From first dose through 10 days post dose.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 5/24
Other Adverse Events (participants affected / at risk) | 17/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=24)
Death (General disorders) | 1 — Not related to study drug
Cardiac arrest (Cardiac disorders) | 1 — Not related to study drug
Necrotising colitis (Gastrointestinal disorders) | 2 — Not related to study drug
Patent ductus arteriosus repair (Surgical and medical procedures) | 1 — Not related to study drug
Septic shock (Infections and infestations) | 1 — Not related to study drug
Renal failure acute (Renal and urinary disorders) | 1 — Not related to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=24)
Endocrine disorders Adrenal Insufficiency (Endocrine disorders) | 4 — Not related to study drug
Convulsion (Nervous system disorders) | 3 — Not related to study drug
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 — Not related to study drug
Other non-serious, infrequent adverse events (General disorders) | 7 — Not related to study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No